CLINICAL TRIAL: NCT03567499
Title: A Randomised, Double-blind, Placebo Controlled, Repeat-dose, Cross-over Phase I Study to Evaluate the Pro-arrhythmic Potential of GSK3039294 in Healthy Participants
Brief Title: Pro-arrhythmic Potential of GSK3039294 in Healthy Subjects
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The decision to end the study was made for GSK portfolio reasons. No subjects were randomised into the study.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 208741
Record Dates: First submitted 2018-06-13; First posted 2018-06-25 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Amyloidosis
Keywords: Pro-arrhythmic; Holter ECG; SAP; Cardiac telemetry; Benign arrhythmic
MeSH Terms: conditions — Amyloidosis

STUDY DESIGN:
Intervention Model Description: This study will consist of two parts, Part A and a conditional Part B. Part A is designed as a randomized double-blinded, 3 period, placebo-controlled, repeat-dose, cross-over study. The decision to initiate Part B will be made based on an evaluation of data from Part A which will include an overall assessment of safety, PK and PD. Part B will also employ a randomized, double-blind, repeat dose, cross-over study design and will follow the same assessments and procedures as Part A.
Who Masked: Participant, Investigator
Masking Description: This will be a double-blinded (Sponsor unblinded) study in which the subjects and site staff (Pharmacist unblinded to prepare study drug) will be blinded for the duration of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Part A: Sequence 1 (Experimental): Subjects in sequence 1 will receive matching placebo in period 1 followed by GSK3039294 200 milligrams (mg) in Period 2 followed by GSK3039294 600 mg in Period 3 once daily orally. There will be a minimum of 7-day washout period between each treatment session. Each treatment session will consist of 7 days of dosing.
  Interventions: Drug: GSK3039294; Drug: Placebo
- Part A:Sequence 2 (Experimental): Subjects in sequence 2 will receive GSK3039294 600 mg in period 1 followed by matching placebo in Period 2 followed by GSK3039294 200 mg in Period 3 once daily orally. There will be a minimum of 7-day washout period between each treatment session. Each treatment session will consist of 7 days of dosing.
  Interventions: Drug: GSK3039294; Drug: Placebo
- Part A: Sequence 3 (Experimental): Subjects in sequence 3 will receive GSK3039294 200 mg in period 1 followed by GSK3039294 600 mg in Period 2 followed by matching placebo in Period 3 once daily orally. There will be a minimum of 7-day washout period between each treatment session. Each treatment session
  Interventions: Drug: GSK3039294; Drug: Placebo
- Part A: Sequence 4 (Experimental): Subjects in sequence 4 will receive GSK3039294 600 mg in period 1 followed by GSK3039294 200 mg in Period 2 followed by matching placebo in Period 3 once daily orally. There will be a minimum of 7-day washout period between each treatment session. Each treatment session will consist of 7 days of dosing.
  Interventions: Drug: GSK3039294; Drug: Placebo
- Part A: Sequence 5 (Experimental): Subjects in sequence 5 will receive GSK3039294 200 mg in period 1 followed by matching placebo in Period 2 followed by GSK3039294 600 mg in Period 3 once daily orally. There will be a minimum of 7-day washout period between each treatment session. Each treatment session will consist of 7 days of dosing.
  Interventions: Drug: GSK3039294; Drug: Placebo
- Part A: Sequence 6 (Experimental): Subjects in sequence 6 will receive matching placebo in period 1 followed by GSK3039294 600 mg in Period 2 followed by GSK3039294 200 mg in Period 3 once daily orally. There will be a minimum of 7-day washout period between each treatment session. Each treatment session will consist of 7 days of dosing.
  Interventions: Drug: GSK3039294; Drug: Placebo
- Part B: Sequence 1 (Experimental): Subjects in sequence 1 will receive matching placebo in period 1 followed by GSK3039294 (dose level to be decided on results of Part 1) in Period 2 once daily orally. There will be a minimum of 7-day washout period between each treatment session. Each treatment session will consist of 7 days of dosing.
  Interventions: Drug: GSK3039294; Drug: Placebo
- Part B: Sequence 2 (Experimental): Subjects in sequence 2 will receive GSK3039294 (dose level to be decided on results of Part 1) in period 1 followed by matching placebo in Period 2 once daily orally. There will be a minimum of 7-day washout period between each treatment session. Each treatment session will consist of 7 days of dosing
  Interventions: Drug: GSK3039294; Drug: Placebo

INTERVENTIONS:
Drug: GSK3039294 — GSK3039294 capsules will be available with a dose strength of 100 mg and 200 mg to be taken as single or multiple capsules orally along with water depending on the dosage required.
Drug: Placebo — Matching placebo capsules to match active 100 mg and 200 mg dose strength will be available and to be taken as single or multiple capsules orally along with water depending on the number of active capsules to blind.

SUMMARY:
GSK3039294 has been developed to offer an orally available alternative to parenteral GSK2315698 (miridesap) for plasma serum amyloid P component (SAP) depletion prior to and following use of anti-SAP Monoclonal Antibody (mAb) in the treatment of systemic amyloidosis. The primary objectives of the study are to assess the cardiac arrhythmic potential of GSK3039294 and evaluate safety and tolerability of repeat doses of GSK3039294, in healthy subjects relative to placebo for the same duration. This study will consist of two parts, Part A and a conditional Part B. Part A is designed as a randomized double-blinded, 3 period, placebo-controlled, repeat-dose, crossover study. The decision to initiate Part B will be based on an evaluation of data from Part A, which will include an overall assessment of safety, pharmacokinetics (PK) and pharmacodynamics (PD). In Part A, there will be three treatment periods with 7 days of dosing in each and minimum 7-day washout period between each treatment session. Each subject will receive two dose levels of GSK3039294 and placebo. In Part B, there will be two treatment periods with 7 days of dosing in each and minimum 7-day washout period. Each subject will receive one dose level of GSK3039294 and placebo. In Part A, approximately 48 subjects will be recruited for an estimated total of 36 completers. In Part B, approximately 32 subjects will be recruited for an estimated total of 24 completers. The study will last up to approximately 10 weeks from screening to follow-up.

ELIGIBILITY:
Eligibility Criteria

Inclusion Criteria:

* 18 to 65 years of age inclusive at the time of signing the informed consent.
* Non-smokers only (defined as a non-smoker during the last 3 months prior to screening).
* Body weight > 50 kilograms and body mass index (BMI) and <=30 kilograms/meter square.
* Male subjects and women of non-child bearing potential only will be eligible.
* Male subjects with female partners of childbearing potential must comply with one of the following contraception requirements from the time of first dose of study medication until completion of the follow-up visit.
* Vasectomy with documentation of azoospermia.
* Male condom plus partner use of one of the contraceptive options: Contraceptive sub dermal implant that meets the effectiveness criteria of a <1% rate of failure per year, as stated in the product label; Intrauterine device or intrauterine system that meets the standard operating procedure (SOP) effectiveness criteria including a <1% rate of failure per year, as stated in the product label; Oral Contraceptive, either combined or progestogen alone; Contraceptive vaginal ring; Occlusive cap (female diaphragm or cervical/vault cap) with a vaginal spermicide (foam, gel, cream or suppository).
* Capable of giving signed informed.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator in consultation with the Medical Monitor if required agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Aspartate aminotransferase, Alanine aminotransferase, Alkaline phosphatase and bilirubin <=1.5 ULN (Upper Limit of Normal) (isolated bilirubin >1.5 ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).

Exclusion Criteria:

* History or presence of/significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study treatment; or interfering with the interpretation of data.
* Clinically significant blood pressure as determined by the investigator.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* QT interval corrected for heart rate according to Fridericia's formula (QTcF)>450 milliseconds.
* Screening 12-lead ECG with any of the following: second/third degree atrioventricular block (AVB); significant pathological Q-waves (defined as Q-wave > 40 milliseconds or depth greater than 0.4-0.5 millivolts); ventricular pre-excitation; complete left bundle branch block (LBBB); bradycardia as defined by sinus rate <= 35 beats per minute (BPM).
* Any clinically relevant abnormality on the screening medical assessment laboratory examination or ECG.
* A personal history of corrected QT interval (QTc) prolongation, symptomatic cardiac arrhythmias or cardiac arrest.
* Sinus bradycardia <= 35 BPM or junctional arrhythmia > 60 BPM for 10 seconds or longer on run-in Holter or pre-dose inpatient telemetry.
* Non-sustained supraventricular tachycardia (NSVT) or more than 30 Ventricular Premature Depolarization (VPD)/hour on run-in Holter or pre-dose inpatient telemetry.
* Atrial tachycardia > 100 BPM for 3 seconds or longer or more than 40 Atrial Premature Depolarization (APD)/hour on run-in Holter or pre-dose inpatient telemetry.
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GlaxoSmithKline (GSK) Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* Participation in the study would result in loss of blood or blood products in excess of 500 milliliters within 56-day period.
* Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Presence of Hepatitis B surface antigen (HBsAg) at screening Positive Hepatitis C antibody test result at screening.
* Positive Hepatitis C Ribonucleic acid (RNA) test result at screening or within 3 months prior to first dose of study treatment.
* Positive pre-study drug/alcohol screen.
* Positive human immunodeficiency virus (HIV) antibody test.
* Regular use of known drugs of abuse.
* Regular alcohol consumption within six months prior to the study defined as: For United Kingdom (UK) sites an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 grams of alcohol: a half-pint (equivalent to 240 milliliters) of beer, one glass (125 milliliters) of wine or one (25 milliliters) measure of spirits.
* Urinary cotinine levels indicative of smoking/history/regular use of tobacco/nicotine-containing products within 3 months prior to screening.
* Sensitivity to heparin or heparin-induced thrombocytopenia.
* Sensitivity to any of the study treatments, or components thereof, or drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07-12 (Estimated); Primary Completion 2019-05-03 (Estimated); Study Completion 2019-05-03 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with benign arrhythmic events measured by Holter Electrocardiogram (ECG): Part A | Up to 44 days
  Benign arrhythmia is defined as one of the following events: atrial fibrillation, supraventricular arrhythmia, ectopic atrial rhythm, ventricular trigeminy, non-sustained ventricular tachycardia, junctional rhythm, accelerated idioventricular rhythm, sinus pause > 3 seconds that are of no clinical significance. Benign arrhythmic events as measured by Holter ECG will be presented,
Number of subjects with benign arrhythmic events measured by Holter ECG: Part B | Up to 27 days
  Benign arrhythmia is defined as one of the following events: atrial fibrillation, supraventricular arrhythmia, ectopic atrial rhythm, ventricular trigeminy, non-sustained ventricular tachycardia, junctional rhythm, accelerated idioventricular rhythm, sinus pause > 3 seconds that are of no clinical significance. Benign arrhythmic events as measured by Holter ECG will be presented,
Number of subjects with benign arrhythmic events as measured by cardiac telemetry: Part A | Up to 38 days
  Benign arrhythmia is defined as one of the following events: atrial fibrillation, supraventricular arrhythmia, ectopic atrial rhythm, ventricular trigeminy, non-sustained ventricular tachycardia, junctional rhythm, accelerated idioventricular rhythm, sinus pause > 3 seconds that are of no clinical significance. Benign arrhythmic events as measured by cardiac telemetry will be presented.
Number of subjects with benign arrhythmic events as measured by cardiac telemetry: Part B | Up to 23 days
  Benign arrhythmia is defined as one of the following events: atrial fibrillation, supraventricular arrhythmia, ectopic atrial rhythm, ventricular trigeminy, non-sustained ventricular tachycardia, junctional rhythm, accelerated idioventricular rhythm, sinus pause > 3 seconds that are of no clinical significance. Benign arrhythmic events as measured by cardiac telemetry will be presented.
Number of subjects with adverse events (AE) and serious adverse events (SAE): Part A | Up to 58 days
  AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect or is medically significant.
Number of subjects with AE and SAE: Part B | Up to 41 days
  AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect or is medically significant.
Number of subjects with abnormal hematology parameters: Part A | Up to 49 days
  Blood samples will be collected for assessment of hematology parameters including platelet count, red blood cell count (RBC), hemoglobin, hematocrit, mean corpuscular volume, mean corpuscular hemoglobin, percentage of reticulocytes, neutrophils, lymphocytes, monocytes, eosinophil's and basophils.
Number of subjects with abnormal hematology parameters: Part B | Up to 35 days
  Blood samples will be collected for assessment of hematology parameters including platelet count, RBC, hemoglobin, hematocrit, mean corpuscular volume, mean corpuscular hemoglobin, percentage of reticulocytes, neutrophils, lymphocytes, monocytes, eosinophil's and basophils.
Number of subjects with abnormal clinical chemistry parameters: Part A | Up to 49 days
  Blood samples will be collected for the assessment of clinical chemistry parameters blood urea nitrogen, creatinine, glucose fasting, potassium, sodium, calcium, aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, total and direct bilirubin and total protein.
Number of subjects with abnormal clinical chemistry parameters: Part B | Up to 35 days
  Blood samples will be collected for the assessment of clinical chemistry parameters blood urea nitrogen, creatinine, glucose fasting, potassium, sodium, calcium, aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, total and direct bilirubin and total protein.
Number of subjects with abnormal urinalysis parameters: Part A | Up to 49 days
  Routine urinalysis will be performed for parameters specific gravity, potential of hydrogen (pH), glucose, protein, blood, ketones, bilirubin, urobilinogen, nitrite, leukocyte esterase by dipstick method and microscopic examination (if blood protein is abnormal).
Number of subjects with abnormal urinalysis parameters: Part B | Up to 35 days
  Routine urinalysis will be performed for parameters specific gravity, pH, glucose, protein, blood, ketones, bilirubin, urobilinogen, nitrite, leukocyte esterase by dipstick method and microscopic examination (if blood protein is abnormal).
Number of subjects with abnormal results on core urine monitoring: Part A | Up to 52 days
  Core urine monitoring will be performed for parameters Spot Urine Protein Creatinine (UPC) ratio and urine pH using a pH meter. Samples for urine pH to be taken in the morning.
Number of subjects with abnormal results on core urine monitoring: Part B | Up to 44 days
  Core urine monitoring will be performed for parameters Spot UPC) ratio and urine pH using a pH meter. Samples for urine pH to be taken in the morning.
Number of subjects with abnormal vital sign parameters: Part A | Up to 58 days
  Vital signs will be measured in a semi-supine position after 5 minutes rest and will include systolic and diastolic blood pressure, and pulse. Blood pressure (systolic and diastolic) and pulse measurements should be preceded by at least 5 minutes of rest for the participant in a quiet setting without distractions.
Number of subjects with abnormal vital sign parameters: Part B | Up to 41 days
  Vital signs will be measured in a semi-supine position after 5 minutes rest and will include systolic and diastolic blood pressure, and pulse. Blood pressure (systolic and diastolic) and pulse measurements should be preceded by at least 5 minutes of rest for the participant in a quiet setting without distractions.
Number of subjects with abnormal 12-lead ECG findings: Part A | Up to 58 days
  ECG's will be obtained as measurements at screening, pre-dose and 1hr post-dose. 12-lead ECGs will be measured in semi-supine position after 5 minutes rest (single electrocardiogram for the presence of any abnormal findings).
Number of subjects with abnormal 12-lead ECG findings: Part B | Up to 41 days
  ECG's will be obtained as measurements at screening, pre-dose and 1hr post-dose. 12-lead ECGs will be measured in semi-supine position after 5 minutes rest (single electrocardiogram for the presence of any abnormal findings).
Number of subjects with abnormal cardiac telemetry findings: Part A | Up to 38 days
  Continuous telemetry will be performed for the assessments of cardiac arrhythmias.
Number of subjects with abnormal cardiac telemetry findings: Part B | Up to 23 days
  Continuous telemetry will be performed for the assessments of cardiac arrhythmias.

SECONDARY OUTCOMES:
Plasma concentration of GSK3039294; Part A | Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16 hours post-dose on Day 1; Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24 hours post-dose on Day 7; Pre-dose on Day 2, 3, 4, 5 and 6 and until follow-up
  Blood samples for PK analysis of GSK3039294 (pro-drug) will be collected at the time points indicated.
Plasma concentration of GSK3039294; Part B | Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16 hours post-dose on Day 1; Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24 hours post-dose on Day 7; Pre-dose on Day 2, 3, 4, 5 and 6 and until follow-up
  Blood samples for PK analysis of GSK3039294 (pro-drug) will be collected at the time points indicated.
Plasma concentration of GSK2315698 (miridesap); Part A | Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16 hours post-dose on Day 1; Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24 hours post-dose on Day 7; Pre-dose on Day 2, 3, 4, 5 and 6 and until follow-up
  Blood samples for PK analysis of GSK2315698 (miridesap) will be collected at the time points indicated.
Plasma concentration of GSK2315698 (miridesap); Part B | Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16 hours post-dose on Day 1; Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24 hours post-dose on Day 7; Pre-dose on Day 2, 3, 4, 5 and 6 and until follow-up
  Blood samples for PK analysis of GSK2315698 (miridesap) will be collected at the time points indicated.
Plasma SAP levels; Part A | Up to 58 days
  Venous blood samples of approximately 4 milliliters will be collected for measurement of SAP. PD effect of repeat doses of GSK3039294 on plasma SAP levels will be recorded.
Plasma SAP levels; Part B | Up to 41 days
  Venous blood samples of approximately 4 milliliters will be collected for measurement of SAP. PD effect of repeat doses of GSK3039294 on plasma SAP levels will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request Site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com